CLINICAL TRIAL: NCT01091831
Title: A Phase 3, Multicentre, Randomized, Controlled Study to Determine the Efficacy and Safety of Cyclophosphamide, Lenalidomide and Dexamethasone (CRD) Versus Melphalan (200 mg/m2) Followed By Stem Cell Transplant In Newly Diagnosed Multiple Myeloma Subjects
Brief Title: Cyclophosphamide, Lenalidomide and Dexamethasone (CRD) Versus Melphalan (200 mg/m2) Followed By Autologous Stem Cell Transplant (ASCT) In Newly Diagnosed Multiple Myeloma Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fondazione EMN Italy Onlus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RV-MM-EMN-441
Record Dates: First submitted 2010-03-22; First posted 2010-03-24 (Estimated); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Lenalidomide; High dose melphalan; Mobilization; CD 34; Newly Diagnosed patients
MeSH Terms: conditions — Multiple Myeloma | interventions — Cyclophosphamide; Lenalidomide; Dexamethasone; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CRD (Active Comparator): Oral therapy with Cyclophosphamide, Lenalidomide and Dexamethasone.
  Interventions: Drug: Cyclophosphamide; Drug: Lenalidomide; Drug: Dexamethasone
- MEL200 (Active Comparator): High dose Melphalan therapy (200 mg/m2) followed by stem cell support for 2 cycles every 4 months (for 1 cycle if at least VGPR was achieved after the 1st MEL200)
  Interventions: Drug: Melphalan

INTERVENTIONS:
Drug: Cyclophosphamide — Cyclophosphamide will be given orally at the dose of 300 mg/m2 on days 1, 8, 15 for 6 cycles every 28 days
  Arms: CRD
Drug: Lenalidomide — Lenalidomide will be given orally at the dose of 25 mg/d for 21 days followed by a 7 days rest period (day 22 to 28)for 6 cycles every 28 days
  Arms: CRD
Drug: Dexamethasone — Dexamethasone will be given orally at the dose of 40 mg on days 1, 8, 15, 22 for 6 cycles every 28 days
  Arms: CRD
Drug: Melphalan — Melphalan will be given iv at the dose of 200 mg/m2 for 1 day followed by stem cell support. The second MEL200 was performed 120 days after the first if ≤ PR was achieved after the 1st MEL200.
  Arms: MEL200

SUMMARY:
This is a multicenter, randomized, open label study designed to compare the efficacy and safety of lenalidomide with low-dose alkylating agents versus high-dose melphalan followed by stem cell support in newly diagnosed symptomatic MM patients who are 65 years of age or younger.

ELIGIBILITY:
Inclusion Criteria:

Patient is, in the investigator(s) opinion, willing and able to comply with the protocol requirements.

* Patient has given voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care.
* Patient is 65 years old or younger at the time of signing the informed consent
* Women of child-bearing potential must agree to use 2 methods of contraception: 1 effective (for example hormonal or tubal ligation) and 1 barrier (for example latex condom, diaphragm) for at least 4 weeks before starting the therapy, during the Treatment Period, and for 4 weeks after the last dose of lenalidomide
* Male patient agrees to use an acceptable method for contraception (i.e., condom or abstinence) during study drug therapy (including dose interruption) and for 4 weeks after discontinuation of lenalidomide therapy.
* Negative serum beta-human chorionic gonadotropin ( beta-HCG) pregnancy test both 24 hours prior to beginning of therapy and then at 4 weeks intervals in women with regular menstrual cycles or every 2 weeks in women with irregular menstrual cycles during study treatment for subjects of childbearing potential
* Patient was diagnosed with symptomatic multiple myeloma based on standard criteria (10), and has measurable disease, defined as follows: any quantifiable serum monoclonal protein value (generally, but not necessarily, greater than 1 g/dL of IgG M-Protein and greater than 0.5 g/dL of IgA M-Protein) and, where applicable, urine light-chain excretion of >200 mg/24 hours; measurable plasmacytoma > 2 cm as determined by clinical examination or applicable radiographs (i.e. MRI, CT-Scan); bone marrow plasma cells >10%.
* Patient has a Karnofsky performance status ≥ 60%.
* Patient has a life-expectancy > 6 months
* Patient has HBV, HCV and HIV negative test.
* Patients must have normal ECG and NYHA ≤ 2; an evaluation of ejection fraction by ECHO or MUGA is optional
* Patients must normal chest X ray; an evaluation of pulmonary function studies on mechanical aspects (FEV1, FVC, etc) and diffusion capacity (DLCO) is optional.
* Patient has the following laboratory values within 14 days before Baseline (day 1 of the Cycle 1):

  * Platelet count ≥ 75 x 109/L without transfusion support within 7 days before the test.
  * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L without the use of growth factors.
  * Corrected serum calcium ≤ 14 mg/dL (3.5 mmol/L).
  * Aspartate transaminase (AST): ≤ 2.5 x the upper limit of normal (ULN).
  * Alanine transaminase (ALT): ≤ 2.5 x the ULN.
  * Total bilirubin: ≤ 1.5 x the ULN.
  * Calculated or measured creatinine clearance: ≥ 20 mL/minute
  * Patient has a baseline bone marrow sample available for cytogenetics, that will be processed and eventually centralized.

Exclusion Criteria:

* Previous treatment with anti-myeloma therapy (does not include radiotherapy, bisphosphonates, or a single short course of steroid; < to the equivalent of dexamethasone 40 mg/day for 4 days).
* Any serious medical condition, including the presence of laboratory abnormalities, which places the subject at an unacceptable risk if he or she participates in this study or confounds the experimental ability to interpret data from the study.
* Pregnant or lactating women. A serum β-hCG pregnancy test must be performed at the Screening visit, for female patients of child-bearing potential. If the test is positive, the patient must be excluded from the study. Confirmation that the patient is not pregnant must be established by a negative serum or urinary pregnancy test with the result obtained 1 day prior to the Baseline visit (or the day of the visit if results are available before drug delivery). A pregnancy test is not required for naturally post-menopausal women (who have not had menses at any time in the preceding 24 consecutive months) or surgically sterilised women (hysterectomy, bilateral ovariectomy, bilateral salpingectomy);
* Prior history of malignancies, other than multiple myeloma, unless the subject has been free of the disease for ≥ 3 years. Exceptions include the following: basal cell carcinoma of the skin, squamous cell carcinoma of the skin, carcinoma in situ of the cervix, carcinoma in situ of the breast, incidental histologic finding of prostate cancer (TNM stage of T1a or T1b)
* Patients previously diagnosed as bearing deep venous thrombosis or arterial thromboembolic event within the latest 12 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 389 (Actual)
Dates: Start 2009-07 (Actual); Primary Completion 2021-09 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Progression free survival | 5 years

SECONDARY OUTCOMES:
Overall survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Gay, MD, Principal Investigator — Division of Hematology - University of Torino - A.O.U. Città della Salute e della Scienza di Torino - Torino - Italy
Locations (1):
- Division of Hematology, A.O.U. Città della Salute e della Scienza di Torino, Torino, Italy

REFERENCES:
- [Derived] Montefusco V, Gay F, Spada S, De Paoli L, Di Raimondo F, Ribolla R, Musolino C, Patriarca F, Musto P, Galieni P, Ballanti S, Nozzoli C, Cascavilla N, Ben-Yehuda D, Nagler A, Hajek R, Offidani M, Liberati AM, Sonneveld P, Cavo M, Corradini P, Boccadoro M. Outcome of paraosseous extra-medullary disease in newly diagnosed multiple myeloma patients treated with new drugs. Haematologica. 2020 Jan;105(1):193-200. doi: 10.3324/haematol.2019.219139. Epub 2019 Jun 20. PMID 31221778
- [Derived] Gambella M, Omede P, Spada S, Muccio VE, Gilestro M, Saraci E, Grammatico S, Larocca A, Conticello C, Bernardini A, Gamberi B, Troia R, Liberati AM, Offidani M, Rocci A, Palumbo A, Cavo M, Sonneveld P, Boccadoro M, Oliva S. Minimal residual disease by flow cytometry and allelic-specific oligonucleotide real-time quantitative polymerase chain reaction in patients with myeloma receiving lenalidomide maintenance: A pooled analysis. Cancer. 2019 Mar 1;125(5):750-760. doi: 10.1002/cncr.31854. Epub 2018 Dec 18. PMID 30561775
- [Derived] Gay F, Oliva S, Petrucci MT, Conticello C, Catalano L, Corradini P, Siniscalchi A, Magarotto V, Pour L, Carella A, Malfitano A, Petro D, Evangelista A, Spada S, Pescosta N, Omede P, Campbell P, Liberati AM, Offidani M, Ria R, Pulini S, Patriarca F, Hajek R, Spencer A, Boccadoro M, Palumbo A. Chemotherapy plus lenalidomide versus autologous transplantation, followed by lenalidomide plus prednisone versus lenalidomide maintenance, in patients with multiple myeloma: a randomised, multicentre, phase 3 trial. Lancet Oncol. 2015 Dec;16(16):1617-29. doi: 10.1016/S1470-2045(15)00389-7. Epub 2015 Nov 17. PMID 26596670